CLINICAL TRIAL: NCT06033833
Title: A Long-term Extension Study to Evaluate the Long-term Safety, Tolerability, and Efficacy of Subcutaneous Amlitelimab in Adult Participants With Moderate-to-severe Asthma Who Completed Treatment Period of Previous Amlitelimab Asthma Clinical Study
Brief Title: Long-term Safety and Efficacy Evaluation of Subcutaneous Amlitelimab in Adult Participants With Moderate-to-severe Asthma Who Completed Treatment Period of Previous Amlitelimab Asthma Clinical Study
Acronym: RIVER-ASTHMA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LTS17510; U1111-1280-5321 (Registry Identifier: ICTRP); 2023-503385-24 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This study will have a double-blind treatment period and an open-label treatment period
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study will have a double-blind treatment period and an open-label treatment period after week 24
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment group 1 (Experimental): Subcutaneous Injection as per protocol
  Interventions: Drug: Amlitelimab
- Treatment group 2 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlitelimab — Injection Solution: by subcutaneous injection (SCI)
  Arms: Treatment group 1
Drug: Placebo — Injection Solution: by subcutaneous injection (SCI)
  Arms: Treatment group 2

SUMMARY:
This is a study of amlitelimab for the treatment of participants with moderate-to-severe asthma. The study will have a double-blind treatment period until Week 24 for each participant and an open-label treatment period where each participant will receive open-label amlitelimab from Week 24 onwards. The purpose of this study is to evaluate long-term safety, tolerability, and efficacy of amlitelimab for the treatment of adult participants with moderate-to-severe asthma who have previously been enrolled and completed the treatment period of the parent study. The study duration will be up to 156 weeks. The treatment duration will be up to 144 weeks. The number of visits will be 18.

DETAILED DESCRIPTION:
The duration of the study for each participant will be up to 156 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate-to-severe asthma who completed the treatment period of the parent study per protocol
* Participants on background dose with medium-to-high doses of ICS therapy (≥500 µg of fluticasone propionate daily or comparable ICS dosage up to a maximum of 2000 µg/day of fluticasone propionate or clinically comparable) in combination with a second or third controller (eg, LABA, LTRA, LAMA, methylxanthines), with or without OCS (up to a maximum of 15 mg prednisone or equivalent daily or 30 mg every other day) as maintained during the parent study in which they participated Note for Japan: participants must be on ≥400 μg of fluticasone propionate daily or equivalent.
* Contraception for male and female participants;

For female participants:

* incapable of becoming pregnant
* not pregnant or breast feeding
* not to donate or cryopreserve eggs for female participants For male participants
* No sperm donation or cryopreserving sperms

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Chronic lung disease other than asthma
* Participants who developed a new medical condition or a change in status of an established medical condition or require a new treatment or medication prior to enrollment, which (per Investigator's medical judgment) would adversely affect the participation in this study or would require permanent IMP discontinuation
* Current smoker or active vaping of any products and/or marijuana smoking
* Prescription drug or substance abuse, including alcohol, considered significant by the Investigator
* Any new development with the participant's disease or condition or any significant laboratory test abnormality during the parent study that, in the opinion of the Investigator, may present an unreasonable risk for the participant
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study
* Individuals accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalized
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures
* Participants are employees of the investigative site or other individuals directly involved in the conduct of the study, or immediate family members of such individuals

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2029-06-25 (Estimated); Study Completion 2029-06-25 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events | From baseline up to Week 156 (EOS of LTS17510)
  Percentage of participants with treatment emergent Adverse Events.

SECONDARY OUTCOMES:
Percentage of participants who experienced adverse events. | From baseline up to Week 156 (End of Study [EOS] of LTS17510)
  Data reported for participants who experienced adverse events of special interest (AESI) and serious adverse events (SAEs).
Annualized rate of severe exacerbation events over treatment period from parent study baseline | From baseline of the parent study up to Week 144 (End of Treatment [EOT] of LTS17510)
  Severe exacerbation events over treatment period from parent study baseline are defined as: Worsening of asthma requiring the use of systemic corticosteroids for ≥3 days (or a single IM or IV injection of corticosteroids) or, in the case of a stable maintenance regimen of oral corticosteroids for the treatment of asthma, a doubling of the dose for 3 or more days; or Hospitalization or emergency room visit or urgent care visit because of asthma, requiring systemic corticosteroids.
Annualized rate of severe exacerbation events over treatment period from LTS17510 study baseline | From baseline of the LTS17510 study Up to Week 144 (EOT of LTS17510)
  Severe exacerbation events over treatment period from LTS17510 study baseline defined as: Worsening of asthma requiring the use of systemic corticosteroids for ≥3 days (or a single IM or IV injection of corticosteroids) or, in the case of a stable maintenance regimen of oral corticosteroids for the treatment of asthma, a doubling of the dose for 3 or more days; or Hospitalization or emergency room visit or urgent care visit because of asthma, requiring systemic corticosteroids.
Time to first exacerbation event from LTS17510 study baseline | From baseline of the LTS17510 study Up to Week 144 (EOT of LTS17510)
Annualized rate of severe asthma exacerbations requiring hospitalization or emergency room or urgent care visit over treatment period from parent study baseline | From baseline of the parent study up to Week 144 (EOT of LTS17510)
  Severe asthma exacerbations are defined as: Worsening of asthma requiring the use of systemic corticosteroids for ≥3 days (or a single IM or IV injection of corticosteroids) or, in the case of a stable maintenance regimen of oral corticosteroids for the treatment of asthma, a doubling of the dose for 3 or more days; or Hospitalization or emergency room visit or urgent care visit because of asthma, requiring systemic corticosteroids.
Annualized rate of severe asthma exacerbations requiring hospitalization or emergency room or urgent care visit over treatment period from LTS17510 study baseline | From baseline of the LTS17510 study up to Week 144 (EOT of LTS17510)
  Severe asthma exacerbations are defined as: Worsening of asthma requiring the use of systemic corticosteroids for ≥3 days (or a single IM or IV injection of corticosteroids) or, in the case of a stable maintenance regimen of oral corticosteroids for the treatment of asthma, a doubling of the dose for 3 or more days; or Hospitalization or emergency room visit or urgent care visit because of asthma, requiring systemic corticosteroids.
Change from parent study baseline in prebronchodilator (BD) and post-BD forced expiratory volume in 1 second (FEV1) at each spirometry endpoint | From baseline of parent study up to week 144 (EOT of LTS17510)
Change from LTS17510 study baseline in pre bronchodilator (BD) and post-BD forced expiratory volume in 1 second (FEV1) at each spirometry endpoint | From baseline of LTS17510 study up to week 144 (EOT of LTS17510)
Change from parent study baseline in pre-BD and post-BD peak expiratory flow [PEF] at each spirometry endpoint | From baseline of parent study up to Week 144 (EOT of LTS17510)
Change from LTS17510 study baseline in pre-BD and post-BD peak expiratory flow [PEF] at each spirometry endpoint | From baseline of LTS17510 study up to Week 144 (EOT of LTS17510)
Change from parent study baseline in Pre-BD and post-BD forced vital capacity [FVC] at each spirometry endpoint | From baseline of parent study up to Week 144 (EOT of LTS17510)
Change from LTS17510 study Baseline in Pre-BD and post-BD forced vital capacity [FVC] at each spirometry endpoint | From baseline of lTS17510 study up to Week 144 (EOT of LTS17510)
Change from parent study baseline in pre-BD and post-BD forced expiratory flow [FEF] 25% to 75%) at each spirometry endpoint | From baseline of parent study up to Week 144 (EOT of LTS17510)
Change from LTS17510 study baseline in pre-BD and post-BD forced expiratory flow [FEF] 25% to 75%) at each spirometry endpoint | From baseline of LTS17510 study up to Week 144 (EOT of LTS17510)
Change from parent study baseline in Asthma Control Questionnaire (ACQ)-5, ACQ-6, and ACQ-7 scores | From parent study baseline up to Week 144 (EOT of LTS17510)
  The ACQ is a validated questionnaire that measures the adequacy of asthma control and any changes in asthma control that may occur spontaneously or as a result of treatment. Each item of the ACQ is measured on a 7-point response scale (0=no impairment, 6=maximum impairment). The ACQ score is the mean of the item responses and ranges from 0 (totally controlled) and 6 (severely uncontrolled).
Change from LTS17510 study baseline in Asthma Control Questionnaire (ACQ)-5, ACQ-6, and ACQ-7 scores | From LTS17510 study baseline up to Week 144 (EOT of LTS17510)
  The ACQ is a validated questionnaire that measures the adequacy of asthma control and any changes in asthma control that may occur spontaneously or as a result of treatment. Each item of the ACQ is measured on a 7-point response scale (0=no impairment, 6=maximum impairment). The ACQ score is the mean of the item responses and ranges from 0 (totally controlled) and 6 (severely uncontrolled).
Change from parent study baseline in Fractional Exhaled Nitric Oxide (FeNO) | From parent study baseline up to Week 144 (EOT of LTS17510)
Change from LTS17510 study baseline in Fractional Exhaled Nitric Oxide (FeNO) | From LTS17510 study baseline up to Week 144 (EOT of LTS17510)
Serum amlitelimab concentrations | From baseline up to Week156 (EOS of LTS17510)
Incidence of anti- amlitelimab antibody positive response | From baseline up to Week 156 (EOS of LTS17510)
Change from parent study baseline and from LTS17510 in Asthma Quality of Life Questionnaire with Standardized Activities (AQLQ [S]) Self-Administered Score | From baseline up to Weeks 144 (EOT of LTS17510)
  The AQLQ(S) was designed as a self-administered participant reported outcome to measure the functional impairments that are most troublesome to adolescents and adults ≥12 years of age as a result of their asthma over the past two weeks. The instrument is comprised of 32 items, each rated on a 7-point Likert scales from 1 to 7.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (68):
- United States (8):
  - Bensch Clinical Research LLC- Site Number : 8400004, Stockton, California
  - Helix Biomedics, LLC - Site Number : 8400029, Boynton Beach, Florida
  - Savin Medical Group - Miami- Site Number : 8400015, Miami, Florida
  - Pines Care Research Center LLC- Site Number : 8400028, Pembroke Pines, Florida
  - Treasure Valley Medical Research- Site Number : 8400031, Boise, Idaho
  - Johns Hopkins University School of Medicine- Site Number : 8400012, Baltimore, Maryland
  - OK Clinical Research, LLC- Site Number : 8400001, Edmond, Oklahoma
  - TTS Research- Site Number : 8400011, Boerne, Texas
- Argentina (9):
  - Investigational Site Number : 0320002, CABA, Buenos Aires
  - Investigational Site Number : 0320008, La Plata, Buenos Aires
  - Investigational Site Number : 0320009, Buenos Aires, Buenos Aires F.D.
  - Investigational Site Number : 0320006, Rosario, Santa Fe Province
  - Investigational Site Number : 0320007, Rosario, Santa Fe Province
  - Investigational Site Number : 0320005, Rosario, Santa Fe Province
  - Investigational Site Number : 0320004, Ciudad Autonoma Bs As
  - Investigational Site Number : 0320003, Ciudad Autonoma Buenos Aires
  - Investigational Site Number : 0320001, Ciudad Autonoma Buenos Aires
- Brazil (7):
  - Centro de Diagnostico e Pesquisa da Osteoporose do Espirito Santo- Site Number : 0760002, Vitória, Espírito Santo
  - Proar- Site Number : 0760004, Salvador, Estado de Bahia
  - Instituto Méderi de Pesquisa e Saúde- Site Number : 0760001, Passo Fundo, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre- Site Number : 0760007, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS- Site Number : 0760006, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas de Sao Paulo- Site Number : 0760008, São Paulo, São Paulo
  - Clínica de Alergia Martti Antila- Site Number : 0760003, Sorocaba
- Canada (2):
  - Investigational Site Number : 1240008, Ottawa, Ontario
  - Investigational Site Number : 1240007, Trois-Rivières, Quebec
- Chile (5):
  - Investigational Site Number : 1520006, Talca, Maule Region
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520008, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Quillota, Región de Valparaíso
- Hungary (4):
  - Investigational Site Number : 3480009, Edelény
  - Investigational Site Number : 3480011, Gödöllö
  - Investigational Site Number : 3480006, Püspökladány
  - Investigational Site Number : 3480012, Százhalombatta
- Italy (3):
  - Investigational Site Number : 3800003, Rome, Roma
  - Investigational Site Number : 3800004, Naples
  - Investigational Site Number : 3800001, Verona
- Japan (5):
  - Investigational Site Number : 3920010, Sakai, Osaka
  - Investigational Site Number : 3920005, Chuo-ku, Tokyo
  - Investigational Site Number : 3920004, Chuo-ku, Tokyo
  - Investigational Site Number : 3920001, Shinagawa-ku, Tokyo
  - Investigational Site Number : 3920019, Hiroshima
- Mexico (4):
  - Investigational Site Number : 4840001, Guadalajara, Jalisco
  - Investigational Site Number : 4840005, Guadalajara, Jalisco
  - Investigational Site Number : 4840002, Chihuahua City
  - Investigational Site Number : 4840008, Mérida
- Poland (6):
  - Investigational Site Number : 6160001, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160006, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160004, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160003, Elblag
  - Investigational Site Number : 6160002, Gdansk
  - Investigational Site Number : 6160007, Tarnów
- South Africa (4):
  - Investigational Site Number : 7100007, Benoni
  - Investigational Site Number : 7100002, Cape Town
  - Investigational Site Number : 7100001, Cape Town
  - Investigational Site Number : 7100004, Middelburg
- South Korea (5):
  - Investigational Site Number : 4100004, Daegu, Daegu
  - Investigational Site Number : 4100006, Moncton, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100005, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
- Turkey (Türkiye) (5):
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920003, Izmir
  - Investigational Site Number : 7920008, Kayseri
  - Investigational Site Number : 7920005, Kocaeli
  - Investigational Site Number : 7920002, Mersin
- Investigational Site Number : 8260001, Bradford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS17510 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25305&tenant=MT_SNY_9011